CLINICAL TRIAL: NCT02371863
Title: SEP-study; The Assessment of Normal Values in Stress Echocardiographic Parameters in Patients After Successful Mitral Valve Repair for Organic Mitral Valve Regurgitation
Brief Title: Normal Values in Stress Echocardiographic Parameters in Patients After Successful Mitral Valve Repair for Organic MR
Acronym: SEP
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, S.A.J. Chamuleau, MD, PhD, UMC Utrecht
Other Study IDs: NL39865.041.14
Record Dates: First submitted 2014-10-07; First posted 2015-02-26 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Heart Valve Diseases; Mitral Valve Insufficiency; Heart; Dysfunction Postoperative, Cardiac Surgery; Heart; Disease, Mitral(Valve); Diseases of Mitral Valve
MeSH Terms: conditions — Heart Valve Diseases; Mitral Valve Insufficiency; Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Surgical treatment is the only approach with potentially defined clinical success for organic mitral valve (MV) regurgitation. Recurrent or persistent complaints after initial successful MV repair is a clinical challenge in current practice. Especially when echo parameters at rest are within or near normal ranges and patients presenting disproportionately symptomatic in relation to the observed results. However, while MV regurgitation is a hemodynamic disease, currently used 2-dimensional (2D) transthoracic echocardiography (TTE) at rest lacks information about hemodynamic changes. Physical stress echocardiography is a promising technique to complement nowadays rest TTE in order to improve interpretation of hemodynamic changes. However, normal values for exercise echo are lacking in this postoperative patients cohort. A prospective, observational trial to determine normal values in stress echocardiographic parameters in asymptomatic patients after successful MV repair for organic MV regurgitation, is therefore highly needed.

Purpose of the SEP- study is to determine normal values in stress echocardiographic parameters in asymptomatic patients at least 6 months after successful MV repair for organic MV regurgitation. These normal values for stress echo are of utmost importance to correctly and accurate interpret stress echo results during postoperative follow-up and to improve clinical decision making in patients post MV repair.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Male or female from all ethnicities;
* At least 6 months post successful, isolated MV repair. S
* Asymptomatic

Exclusion Criteria:

* Pulmonary hypertension >50 mmHg at rest;
* Atrial fibrillation (AF) at time of study related stress echo test;
* Known contraindication or incapability to perform peak exercise or inability to perform physical stress testing;
* LVEF <45%;
* NYHA class II and more.
* Other heart valve disease of more than mild severity;
* Concomitant surgery during MV repair, e.g. MAZE, TVP procedure;
* Prior heart valve surgery;
* Congenital heart disease;
* Disabling comorbidity, e.g. chronic obstructive pulmonary disease (COPD);
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 Asymptomatic patients (≥18 years) at least 6 months after successful MV repair. Patients will have a LVEF ≥45%, and were initially operated based on organic MV regurgitation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Echocardiographic parameter: Peak mitral valve mean gradient (mmHg) | at least 6 months after successful MV repair
  Echocardiographic measured mitral valve mean gradient at peak physical exercise
Echocardiographic parameter: Peak systolic pulmonary artery pressure (sPAP, mmHg) | at least 6 months after successful MV repair
  Echocardiographic measured sPAP at peak physical exercise
Echocardiographic parameter: Increase in mitral valve regurgitation grade (grade 0-4, according to ESC guidelines) | at least 6 months after successful MV repair
  Echocardiographic measured increase in mitral valve regurgitation at peak physical exercise during physical stress echo, compared to rest echo. Grading of mitral regurgitation will be performed according to the ESC guidelines.

SECONDARY OUTCOMES:
Echocardiographic parameter: Left ventricular function (LVF, quality description) | at least 6 months after successful MV repair
  Echocardiographic measured LVF quality at rest and peak physical exercise
Echocardiographic parameter: Mitral valve area (MVA, cm2) | at least 6 months after successful MV repair
  Echocardiographic measured MVA at rest and peak physical exercise
Echocardiographic parameter: Peak mitral valve peak gradient (mmHg) | at least 6 months after successful MV repair
  Echocardiographic measured mitral valve peak gradient at peak physical exercise

CONTACTS AND LOCATIONS:
Overall Officials: Steven AJ Chamuleau, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht (UMC Utrecht), Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Jansen R, Urgel K, Cramer MJ, van Aarnhem EEHL, Zwetsloot PPM, Doevendans PA, Kluin J, Chamuleau SAJ. Reference Values for Physical Stress Echocardiography in Asymptomatic Patients after Mitral Valve Repair. Front Surg. 2018 Feb 19;5:6. doi: 10.3389/fsurg.2018.00006. eCollection 2018. PMID 29516004